CLINICAL TRIAL: NCT06076382
Title: A Prospective Randomized Controlled Study Protocol Between Endoscopic Ultrasound Guided Colorectal ESD and Traditional Colorectal ESD Surgery
Brief Title: Endoscopic Ultrasound Guided Colorectal ESD and Traditional Colorectal ESD Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jilin University (Other)
Responsible Party: Principal Investigator, Dong Yang, Assisted Investigator, Jilin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 130026
Record Dates: First submitted 2023-09-24; First posted 2023-10-10 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Endoscopic Submucosal Dissection(ESD) Surgery
Keywords: colorectal; Endoscopic submucosal dissection; ultrasound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the endoscopic ultrasound guided colorectal ESD surgery group (Experimental): The experimental group first underwent endoscopic ultrasound examination, with a small ultrasound probe inserted into the intestinal cavity through the biopsy port. Then undergo the colorectal ESD surgery.
  Interventions: Procedure: endoscopic ultrasound guided colorectal ESD surgery
- the traditional colorectal ESD surgery group (Active Comparator): the traditional colorectal ESD surgery
  Interventions: Procedure: the traditional colorectal ESD surgery

INTERVENTIONS:
Procedure: endoscopic ultrasound guided colorectal ESD surgery — The experimental group first underwent endoscopic ultrasound examination, with a small ultrasound probe inserted into the intestinal cavity through the biopsy port. After water injection, the lesion was scanned and (1) the direction of gravity was determined. (2) fibrosis/infiltration under the mucosa, and the fibrosis was divided into F0 (no fibrosis), F1 (cold fibrosis), or F2 (severe fibrosis). (3) The lesion was divided into nine compartments. Mark submucosal fibrosis/infiltration sites, according to nine compartments. (4) Based on the results of endoscopic ultrasound scanning of the lesion, the surgeon draw up surgical approach and perform injection and dissection.
  Arms: the endoscopic ultrasound guided colorectal ESD surgery group
Procedure: the traditional colorectal ESD surgery — The control group underwent injection and dissection directly.
  Arms: the traditional colorectal ESD surgery group

SUMMARY:
A prospective randomized controlled study protocol between endoscopic ultrasound guided colorectal ESD and traditional colorectal ESD surgery

DETAILED DESCRIPTION:
This study compare and analyze the efficiency of endoscopic ultrasound guided colorectal ESD surgery with traditional colorectal ESD surgery, in order to guide colorectal ESD operations.

ELIGIBILITY:
Inclusion Criteria:

* Cases in our hospital who require colorectal ESD surgery
* Colorectal lesions（laterally spreading tumor）.

Exclusion Criteria:

* Laterally spreading tumor but not nodular mixed type(LST-G-M)
* Patients who have participated or are currently participating in other clinical trials within the first 4 weeks of enrollment;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2024-12-28 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
operating time | During surgery
  from the injection to the end of dissection （minutes）
Measure the area of the lesion | During surgery
  Measure the length and diameter of the lesion

SECONDARY OUTCOMES:
Number of propria muscle layer injuries during surgery | During surgery
  record the points of propria muscle layer injuries during surgery
Time to first fluid diet | one week after surgery
  Postoperative recovery: record the first time of fluid diet
Complete resection rate | 1 year
  record the number of complete resection cases

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No